CLINICAL TRIAL: NCT04768413
Title: Evaluation of a Non-face to Face Multidisciplinary Health Care Model in a Population With Rheumatoid Arthritis Highly Vulnerable to the 2019 Novel Coronavirus Disease
Brief Title: Evaluation of a Non-face to Face Multidisciplinary Health Care Model in a Population With Rheumatoid Arthritis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Fundación Universitaria de Ciencias de la Salud (Other)
Collaborators: Biomab I.P.S. Centro de Atencion Integral en Artritis Reumatoide (Other)
Responsible Party: Sponsor
Other Study IDs: 5171
Record Dates: First submitted 2020-11-27; First posted 2021-02-24 (Actual); Last update posted 2021-02-24 (Actual); Status verified 2021-02

CONDITIONS: Rheumatoid Arthritis
Keywords: Rheumatoid Arthritis; Telemedicine; Telehealth; COVID-19; Disease Activity; Outcomes research
MeSH Terms: conditions — Arthritis, Rheumatoid; COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 9 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group A: A group of patients who have voluntarily adhered to the clinic's tele-assisted consultation and who receive remote, multidisciplinary team care without requiring physical displacement.
  Interventions: Other: Teleconsultation either by phone or by computer consultation. Quantitative and qualitative approaches to analysis
- Group B: Group of patients who wish to continue with the usual face-to-face consultation, since for these patient's isolation measures allow trips to the care centers and who receive care from a multidisciplinary team on a regular basis.
  Interventions: Other: Care modalities. Quantitative and qualitative approaches to analysis

INTERVENTIONS:
Other: Teleconsultation either by phone or by computer consultation. Quantitative and qualitative approaches to analysis — A group of patients who have voluntarily adhered to the clinic's tele-assisted consultation and who receive remote, multidisciplinary team care without requiring physical displacement.
  Groups: Group A
Other: Care modalities. Quantitative and qualitative approaches to analysis — Group of patients who wish to continue with the usual face-to-face consultation, since for these patient's isolation measures allow trips to the care centers and who receive care from a multidisciplinary team on a regular basis.
  Groups: Group B

SUMMARY:
This research work proposes the evaluation of the implementation of a tele-orientation program and tele-consultation to the adult population with RA attended at a specialized rheumatology center in Bogota, Colombia, over a period of three months, by means of a observational, analytical, cohort, prospective study that will include mixed methods for collecting information (quantitative and qualitative)

DETAILED DESCRIPTION:
The evaluation of the priority implementation of a non-face-to-face multidisciplinary health care model is justified in a population highly vulnerable to COVID 19, with Rheumatoid arthritis (RA) in a health emergency situation and in turn seeking to promote its well-being, taking into account the importance of interdisciplinary follow-up to strengthen self-care, avoid deterioration, hospital admissions and improve therapeutic adherence. This research work proposes the evaluation of the implementation of a tele-orientation program and tele-consultation to the adult population with RA attended at a specialized rheumatology center in Bogota, Colombia, over a period of three months, by means of a observational, analytical, cohort, prospective study that will include mixed methods for collecting information (quantitative and qualitative). The qualitative methods will include interviews with a subgroup of patients attending by the two models and with the professionals who care for them, with the aim of knowing the experiences and perceptions of both the patients and the professionals.

The impact that the project seeks is focused on evaluating the program's contribution to the control of RA symptoms and inflammation, avoiding progressive structural damage.

On the other hand, elements will be provided to advance towards telehealth educational interventions and their effect in improving the therapeutic adherence of patients with RA, as well as avoiding their displacement, maintaining quarantine measures and stimulating necessary self-care measures in search of mitigate the COVID-19 pandemic and counteract the spread of the severe acute respiratory syndrome coronavirus 2, particularly in this susceptible risk group.

Finally, this study will provide information on the characteristics of RA patients who choose telemedicine compared to face-to-face care when both are offered as usual care options during an unprecedented situation such as the COVID-19 pandemic. For this reason, the possibility of replication at the national level from the planning of telemedicine programs in rheumatology will be essential for contributing to the reduction of epidemiological indicators against contagion by coronavirus and the use of hospital service

ELIGIBILITY:
Inclusion Criteria:

* Quantitative and qualitative approach. Patients over 18 years of age with confirmed diagnosis of rheumatoid arthritis International Classification of Diseases: M069, M059, M060, treated at a reference center for these pathologies in the city of Bogotá.
* Quantitative approach Patients with access to information and communication technologies
* Qualitative approach: Patients seen in the teleconsultation modality on at least two occasions.
* Qualitative approach: Patients attended in the face-to-face consultation modality on at least two occasions.
* Qualitative approach: Health professionals who have carried out at least 25 teleconsultations directed at patients with rheumatoid arthritis in a reference center for these pathologies in the city of Bogotá.

Exclusion Criteria:

* Patients who due to their cognitive conditions do not have the ability to provide reliable information necessary for the development of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Rheumatoid Arthritis patients regularly followed in a in a specialized rheumatology center in Bogota, Colombia
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2020-06-01 (Actual); Primary Completion 2021-04-30 (Estimated); Study Completion 2021-06-30 (Estimated)

PRIMARY OUTCOMES:
Evaluation of the implementation of a non-face-to-face multidisciplinary consultation model in a population of rheumatoid arthritis | up to Week 12
  Evaluate the implementation of a non-face-to-face multidisciplinary consultation model in a population with rheumatoid arthritis, highly vulnerable to severe acute respiratory syndrome coronavirus 2 [coronavirus disease (COVID-19)] during a health emergency situation and evaluation of the effectiveness of their results.

SECONDARY OUTCOMES:
Epidemiological characterization | up to Week 12
  Epidemiological characterization of the population evaluated under the multidisciplinary health care model, both in teleconsultation and face-to-face consultation.
Proportion of individuals infected | up to Week 12
  To determine the proportion of individuals infected with severe acute respiratory syndrome coronavirus 2 [coronavirus disease (COVID-19)] in those patients who regularly receive different immunosuppressive medications under the two care models (teleconsultation and face-to-face).
Risk factors for infection | up to Week 12
  Describe the risk factors for severe acute respiratory syndrome coronavirus 2 [coronavirus disease (COVID-19)] infection in the group of patients linked to the teleconsultation model and in those with regular face-to-face care.
Risk factors for hospitalization | up to Week 12
  Describe the risk factors for hospitalization associated with severe acute respiratory syndrome coronavirus 2 [coronavirus disease (COVID-19)] in the group of patients linked to the teleconsultation model and in those with regular face-to-face care.
Risk factors for mortality | up to Week 12
  Describe the risk factors for mortality associated with severe acute respiratory syndrome coronavirus 2 [coronavirus disease (COVID-19)] in the group of patients linked to the teleconsultation model and in those with regular face-to-face care.
Average change from baseline in Disease Activity Score with 28-joint counts [DAS28] in face-to-face consultation group | up to Week 12
  A single score on a continuous scale (0-9.4). The level of disease activity will be interpreted as remission (DAS28 <2.6), low (2.6 ≤ DAS28 < 3.2), moderate (3.2 ≤DAS28≤ 5.1), or high (DAS28 >5.1).
Average change from baseline in Patient Activity Scale scores in both groups tele-assisted consultation and face-to-face consultation | up to Week 12
  The Patient Activity Scale is calculated by multiplying the Health Assessment Questionnaire (HAQ) by 3.33 and then dividing the sum of the visual analogue scale (VAS) pain, Patient global assessment (PtGA), and Health Assessment Questionnaire (HAQ) by 3. Activity will be interpreted as these categories of disease activity: remission ≤0.25, low ≤3.7, moderate <8.0, and high ≥8.0.
Evaluation of participant's pain using visual analogue scale [VAS] in both groups tele-assisted consultation and face-to-face consultation | Baseline, Week 6 and 12
  Paint measurement for any disease state 0-10 centimeters VAS by the patient
Evaluation of the disease activity by Doctor using visual analogue scale [VAS] in both groups tele-assisted consultation and face-to-face consultation | Baseline, Week 6 and 12
  Activity measurement for any disease state 0-10 centimeters VAS by the Doctor
Absolute and percent change in the Health Assessment Questionnaire (HAQ) in both groups tele-assisted consultation and face-to-face consultation | Baseline, Week 6 and 12
  The questionary includes 20 daily life questions, grouped in 8 areas, each one containing two or three questions related to daily life activities. Each question is scored from 0-3. 0 means no disability, 3 score means completely disabled. The average of all responses is done. Average scores from 0-1 represent "mild to moderate difficulty", 1-2 means "moderate to severe disability", 3-2 indicates "severe to very severe disability".
Average change from baseline in European Quality of Life 5 Dimensions (EQ-5D) questionnaire in both groups tele-assisted consultation and face-to-face consultation | up to Week 12
  European Quality of Life 5 Dimensions (EQ-5D) questionnaire is a self-reported health outcome which measures Quality of life (QoL) in five dimensions. An overall score is derived that measures from the least (worst) to the highest score (best). In addition, health state is measured on the vertical Visual Analogue scale (score 0 to 100) with higher scores (better health status).
Evaluation of the level of therapeutic adherence using a specific Scale in both groups tele-assisted consultation and face-to-face consultation | Baseline and week 12.
  The four item MORISKY-GREEN-LEVINE Medication Adherence Scale (MGLS) results in a score ranging from 0 to 4. There are three levels of medication adherence based on this score: high, medium and low adherence with 0, 1-2, and 3-4 points, respectively. A dichotomous definition of adherence based on MGLS will be used with 0 points indicating perfect adherence and 1+ points indicating some level of non-adherence.
Evaluation of the self-care capacity using the Appraisal of Self-care Agency Scale -Revised (ASA-R) in both groups tele-assisted consultation and face-to-face consultation | Baseline and week 12.
  The Appraisal of Self-care Agency Scale -Revised (ASA-R; Sousa et al.) is one of the main instruments to assess self-care capacity. It consists of a total of 15 questions in 3 areas, of which the area lacking self-care agency is reversely coded. Based on a 5-point Likert scale, a higher total score signified a higher level of self-care agency.

OTHER OUTCOMES:
Description of individual experiences of patients: Qualitative data analysis | The moment of the interview (week 12)
  A semi-directed interview will be undertaken with patients with rheumatoid arthritis. The aim will be to obtain a description of their experiences concerning how their health care was developed during the pandemic time and how health-related decisions are made individually considering the interactions with health care professionals in both models face to face and teleconsultation.
Description of individual experiences of health care professionals: Qualitative data analysis | The moment of the interview (week 12)
  Health care professionals will also be interviewed regarding their experiences and needs in rheumatoid arthritis attention based on the two models, in the shared decision-making process and in establishing objective medical decisions.

CONTACTS AND LOCATIONS:
Overall Officials: Adriana Rojas-Villarraga, MD;Rhe, Principal Investigator — FUNDACION UNIVERSITARIA DE CIENCIAS DE LA SALUD
Locations (2):
- Colombia (2):
  - BIOMAP IPS Centro de Atención Integral en Artritis Reumatoide, Bogota, Cundinamarca
  - Colombia Fundación Universitaria de Ciencias de la Salud-FUCS, Bogota, Cundinamarca

IPD SHARING:
Plan to Share IPD: No